CLINICAL TRIAL: NCT06943261
Title: Effects of Task-oriented Training on Visual-motor Integration and Upper Limb Function in Children With Down Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR/AHS/25/ Sajal Waheed
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Down Syndrome
Keywords: Down's syndrome; Visual motor integration; Task-oriented training; Upper limb function
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: A Randomized controlled trial performed in which 28 Down Syndrome children with the age of 6-12 age, will be taken randomly after screening and meeting inclusion criteria. children will be divide in to two groups. Group A (experimental group) will receive task-oriented training of 8 weeks for 30-45 min 3 days a week and (control group) will receive a conventional therapy and game based interventions of 8 weeks for 30-45 min 3 days a week. pre values were take from week 1 and then on week 4 mid values of intervention will be taken and at the end post values of interventions will be taken to measure the effects of both therapies
Who Masked: Participant
Masking Description: participants will get separated treatment protocol and possible effects will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: task oriented training (Experimental): experimental group will receive session of 30 to 45 min of 3 times a week for eight weeks
  Interventions: Other: task oriented training; Other: conventional therapy
- control group : conventional therapy and game based interventions (Active Comparator): control group will receive session of 30 to 45 min of 3 times a week for eight weeks
  Interventions: Other: task oriented training; Other: conventional therapy

INTERVENTIONS:
Other: task oriented training — The 8-week intervention program targets fine motor and functional play skills in children through progressive weekly activities. Week 1 focuses on eye-hand coordination (e.g., stacking blocks, bead stringing), followed by grasp and release control in Week 2 (e.g., object transfer tasks). Week 3 enhances reaching and precision (e.g., targeting and catching), while Week 4 develops bilateral coordination (e.g., buttoning, tearing paper). Week 5 works on visual-motor planning (e.g., drawing, tracing), and Week 6 encourages daily functional play (e.g., pouring, pretend cooking). Week 7 combines skills (e.g., dressing a doll, coin placement), and Week 8 consolidates learning through review and practice of previous tasks.
Other: conventional therapy — The control group will receive standard physical therapy consisting of general exercises aimed at improving overall strength, flexibility, and gross motor skills, without specifically targeting visual-motor integration or fine motor skills. Sessions will also include non-specific recreational activities such as free play or unstructured tasks. The intervention will be conducted three times per week, with each session lasting 45-60 minutes, over a total duration of 8 weeks.

SUMMARY:
The condition known as Down Syndrome (DS) is caused by trisomy 21, or the presence of an extra copy of chromosome 21. DS is the most common survivable autosomal aneuploidy and one of the genetically complicated problem compatible with post-term human survival. Based on current birth prevalence, the prevalence of DS is around 25%-40%. It is one of the most prevalent disease. Visual-motor integration difficulties are common in children with DS, which affects their capacity to synchronize hand movements with vision. This may have an impact on ADLS like writing, eating, grooming. Both delays in motor skills and visual processing might cause difficulties in this domain.

This study will be a randomized controlled trial conducted in spectrum clinic. This study will be completed in time duration of 10 months after approval of synopsis. Non-probability convenience sampling technique will be used and 28 participants will be recruited in study after randomization. Informed consent will be taken from gradians then, the subjects will be divided into two groups and the Group A (Experimental group) will receive task-oriented training 3 times a week which focus on exercises that improve UL function and visual motor coordination and Group B (Control group) will receive general physiotherapy plan and game-based interventions. Poor visual motor skills are one of the inclusion criteria, but significant intellectual disability, prior involvement in related interventions, and untreated medical or psychological conditions are among the exclusion criteria. The data will be assessed at the baseline and after 8th week of treatment. After data collection data will be analyzed by using SPSS version 23.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosed down syndrome patient

  * Both male and female
  * Age range 5 to 12
  * Children who has poor VM skills

Exclusion Criteria:

* • Sever intellectual disability

  * Previous participation in similar interventions
  * Uncontrolled medical or psychiatric conditions
  * Low communication skills

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-06-16 (Estimated)

PRIMARY OUTCOMES:
Jebson Taylor Hand Function Test (JTHFT) | baseline, 4th week,8th week
  ) is a widely used tool for assessing upper limb function in individuals with conditions such as Down syndrome. It evaluates various hand activities, including grasp, manipulation, and coordination, providing valuable insights into the individual's functional abilities and limitations.The Length of the test is 15-45 minutes to complete the JTHFT. JTHFT had moderate to high test-retest reliability and excellent inter-rater reliability (r=0.84 and 0.85, P<0.05) with absent practice effect (P<0.05)
Beery-Buktenica Developmental Test of Visual-Motor Integration (Beery VMI) | baseline, 4th week,8th week
  it is a widely used assessment tool designed to evaluate visual-motor integration skills across various age groups.It takes almost 10 to 15 min to complete the task.The test retest reliability is excellent (0.84-0.88). The Interrater reliability is (0.90-0.98)

CONTACTS AND LOCATIONS:
Overall Officials: Sajal Waheed, MS-PT, Principal Investigator — Riphah International University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thant AA, Wanpen S, Nualnetr N, Puntumetakul R, Chatchawan U, Hla KM, Khin MT. Effects of task-oriented training on upper extremity functional performance in patients with sub-acute stroke: a randomized controlled trial. J Phys Ther Sci. 2019 Jan;31(1):82-87. doi: 10.1589/jpts.31.82. Epub 2019 Jan 29. PMID 30774211